CLINICAL TRIAL: NCT03548961
Title: GI-116: Phase II Study of Organ Preservation in Early Rectal Cancer Patients
Brief Title: Organ Preservation in Early Rectal Cancer Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GI-116; 18-1013 (Other: FCCC)
Record Dates: First submitted 2018-05-25; First posted 2018-06-07 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant chemotherapy (Experimental)
  Interventions: Drug: FOLFOX regimen

INTERVENTIONS:
Drug: FOLFOX regimen — FOLFOX regimen will be administered for 6 cycles. Each cycle is 14 days followed by restaging, local surgery and concurrent chemo radiation therapy

SUMMARY:
This is a single arm phase II study of neoadjuvant chemotherapy followed by local excision and post-operative chemoradiotherapy in patients with early stage, low rectal adenocarcinoma. After completion of pre-treatment tests/procedures (including pelvic MRI/ERUS; MRI is mandatory at baseline and other imaging is encouraged) and confirmation of eligibility, systemic therapy with FOLFOX will be administered for 12 weeks. 2 to 4 weeks after the chemotherapy, restaging of the primary tumor will be done to evaluate response to therapy (Pelvic MRI and /or sigmoidoscopy). Patients with disease progression or inadequate response to chemotherapy to allow local excision will continue with evaluation and treatment per the current standard of care (chemoradiation followed by TME). These patients will be considered failures for the primary endpoint of the study. Patients who respond to the neoadjuvant chemotherapy will proceed with local excision (open, TEMS or TAMIS), 6-12 weeks after the completion of neoadjuvant chemotherapy, followed by 5-FU based chemoradiotherapy 4-12 weeks after local excision. Patients with positive margins at the time of local excision will also be treated as per standard of care and will be considered as failures. Number of patients who can undergo successful local excision with this approach will define the success of the strategy. After chemoradiation therapy post local excision, patients will be followed closely every 3 months for the first 3 years and then every 2 months for the next 2 years (history/physical, CEA and pelvic MRI). Patients who are deemed failures for the primary end-point will be followed as per standard of care, off-study.

ELIGIBILITY:
Inclusion criteria

1. Histologically proven adenocarcinoma of the lower rectum (lower border ≤6 cm from anal verge as assessed by pelvic MRI).
2. Clinical stage T1N0, T2N0, T3N0; high risk T1 and low risk T3 stage patients are also allowed. Clinical staging should be estimated based on the combination of the following assessments: physical exam by the primary surgeon, CT Chest/Abdomen/Pelvis or PET/CT along with Pelvic MRI and Endoscopic Rectal Ultrasound (ERUS). If a pelvic MRI is performed, it is acceptable to perform CT of the chest/abdomen, omitting CT imaging of the pelvis.
3. No prior therapy for rectal cancer
4. Age > 18 years.
5. ECOG performance status 0 or 1
6. Patients must have normal organ and marrow function as defined below

   * Leukocytes > 3,000/mcL
   * Absolute neutrophil count > 1,500/mcL
   * Platelets > 100,000/mcL
   * Total bilirubin < 1.5 times ULN
   * AST/ALT (SGOT/SGPT) < 3 times institutional normal limits
   * Creatinine < 1.5 times ULN OR
   * Creatinine clearance > 60 Ml/min/1.73 m2 for patients with creatinine levels above institutional normal
7. Ability to understand and willingness to sign a written informed consent and HIPAA consent document

Exclusion Criteria:

1. Patients with contraindication to use FOLFOX chemotherapy and pelvic radiation.
2. Low risk T1 tumors that fulfill all of the following - size<4 cm, lack of lymphovascular invasion and well differentiated histology, are excluded
3. High risk T3 tumors that fulfill any of the following - circumferential tumor, extension into mesorectal fascia > 5mm, prediction of positive circumferential resection margin, are also excluded.
4. T4, node positive or advanced rectal adenocarcinoma. Node positivity defined as nodes greater than 1cm in short axis with loss of uniform cortex/fatty hilum
5. Patients receiving other investigational agents
6. Patients who have had chemotherapy (for other malignancies) within 3 years prior to registration
7. Patients with any prior pelvic radiation therapy
8. Prior malignancies requiring systemic therapy within the last 3 years (as prior therapy can increase toxicity of current chemo regimen, those patients should be excluded).
9. History of allergic reactions attributed to compound of similar chemical or biologic composition to the agents used in this study
10. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
11. Known HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with chemotherapeutic drugs. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
12. Pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
number of patients whose tumor can be resected by local excision with negative margins | 3 months
  Patients who undergo neoadjuvant chemotherapy, and are able to achieve a local excision in early stage lower rectal adenocarcinoma with negative margins

SECONDARY OUTCOMES:
Number of patients with improved bowel function in patients treated with organ preserving approach for early stage low rectal cancer before and after therapy | 3 years
  Bowel function will be assessed by Bowel Function Index- Functional Assessment of Chronic Illness Therapy (FACIT) version 4 survey to be completed by patients. The survey measures- Physical well-being, social/family well-being, emotional well-being, functional well-being
Number of patients with improved sexual function treated with organ preserving approach for early stage low rectal cancer before and after therapy | 3 years
  Sexual function in women will be assessed by Female Sexual Function Index (FSFI) 2000 and in men will be assessed by International Index of Erectile Function (IIEF) questionnaire respectively to be completed by patients. The questions ask about the patients' sexual feelings and responses.
Number of patients with improved health-related quality of life treated with organ preserving approach for early stage low rectal cancer before and after therapy | 3 years
  Quality of life will be assessed by Patient Reported Outcome Measurement Information System-10 (PROMIS-10) questionnaire to be completed by patients. This questionnaire will have 10 questions.PROMIS Global-10 allows each of the individual items to be examined separately to provide specific information about perceptions of physical function, pain, fatigue, emotional distress, social health and general perceptions of health.
Overall survival (OS) of patients | 5 years
  OS will be assessed from start of treatment for disease that the patient is still alive
Disease-free survival (DFS) of patients | 5 years
  DFS will be assessed as the length of time that patient survived without any sign of symptoms of that cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided